CLINICAL TRIAL: NCT06122064
Title: Shared Decision-Making Encounter Tool for Adjuvant Treatment of Lung Cancer: Randomized Control Trial
Brief Title: A Tool for Improving the Shared Decision-making Process in Patients With Non-small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-003089; NCI-2023-07463 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-003089 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-10-30; First posted 2023-11-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Videotape Recording; Sound Recordings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (standard of care) (Active Comparator): Patients attend a standard of care visit with their clinician on study.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review; Other: Survey Administration; Other: Video Recording; Other: Audio Recording
- Arm II (standard of care, conversation aid) (Experimental): Patients attend a standard of care visit with the use of the shared decision-making conversation tool by the clinician on study.
  Interventions: Other: Best Practice; Other: Communication Intervention; Other: Electronic Health Record Review; Other: Survey Administration; Other: Video Recording; Other: Audio Recording

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Other: Communication Intervention — Use shared decision-making conversation tool
  Arms: Arm II (standard of care, conversation aid)
Other: Electronic Health Record Review — Ancillary studies
Other: Survey Administration — Ancillary studies
Other: Video Recording — Ancillary studies
Other: Audio Recording — Ancillary studies

SUMMARY:
This clinical trial compares the use of a shared decision-making communication tool during a clinical encounter to standard care for improving the quality of the shared decision-making process among patients with non-small cell lung cancer. Lung cancer patients are faced with many decisions about their treatment options. Studies have found that patients are most satisfied if they perceive an effort by their physician to share decision making and are afforded sufficient time to make their decision. Shared decision-making tools can help physicians guide the conversation, offer tailored estimates of the potential benefits, harms, and practical inconveniences of the available options, and support deliberations that take into account patient biological and biographical circumstances, goals, and priorities. Incorporating a shared decision-making communication tool into standard clinical encounters may improve the shared-decision making process as well as patient satisfaction with their treatment choice.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Encounters where standard of care and the non-small cell lung cancer (NSCLC) choice conversation aid were utilized will have an improvement in the quality of the shared decision-making process over encounters with standard of care alone.

II. Patients with encounters where the NSCLC choice conversation aid was used along with standard of care will have decreased decisional conflict in regard to treatment choice compared to standard of care alone.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients attend a standard of care visit with their clinician on study.

ARM II: Patients attend a standard of care visit with the use of the shared decision-making conversation tool by the clinician on study.

After completion of study intervention, patients are followed up at 2 and 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* CLINICIANS:
* All clinicians within identified departments participating are eligible (doctor of medicine [MD]/doctor of osteopathy [DO], fellows/residents, physician assistant [PA]/nurse practitioner [NP])
* PATIENTS:
* Adult patients (>= 18 years of age)
* Appointments at Mayo Clinic in Rochester
* Non-small cell lung cancer (NSCLC) stage > 1B
* Eligible by their oncologist for adjuvant treatment

Exclusion Criteria:

* Exclude patient with major barriers to provide written informed consent or to participate in shared decision-making (i.e., dementia, severe hearing or visual impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the intervention on implementing shared decision making | Baseline (immediately following appointment); 2 weeks post appointment
  Effectiveness of the intervention will be assessed using the 9-item Shared Decision Making Questionnaire (SDMQ-9) to evaluate standard of care alone versus using the non-small cell lung cancer (NSCLC) conversation aid plus standard of care. The overall score is the sum of the 9 items, where lower values indicate less perceived shared decision making, and higher scores indicate more perceived shared decision making. Self-reported responses from patients and clinicians will also be collected at multiple timepoints throughout the study.
Degree of involvement of patients by the clinician in the shared decision making | Baseline (immediately following appointment); 2 weeks post appointment
  Evaluated using the 12-item "observing patient involvement" (OPTION12) tool, where reviewers will view and score recorded encounters. The survey tool consists of 12 items scored from 0-4, where 0=no effort and 4=exemplary effort.
Provider satisfaction with NSCLC choice conversation aid | After each encounter for the duration of the study, until accrual is reached
  Provider satisfaction with each encounter will be assessed with two questions. The first will be answered using a 5-point Likert scale where 1=Not at all satisfied and 5=Completely satisfied. The second will be answered using a 7-point scale where 1=No, I would strongly recommend against it and 7=Yes, I would strongly recommend it. Higher overall scores indicate higher satisfaction with the intervention.

OTHER OUTCOMES:
Knowledge transfer | Baseline (immediately following appointment); 2 weeks post appointment
  Knowledge transfer will be assessed using 6 questions about treatment options to prevent recurrence of lung cancer. The 6 questions use a response format of "True / False / Do not know". Correct responses will be summed and divided by the total number of questions asked. If a patient answers at least 1 knowledge question then they will be assessed for this outcome, where all missing responses will be coded as incorrect.
Patient satisfaction | Baseline (immediately following appointment); 2 weeks post appointment
  Patient satisfaction with encounter will be assessed with 1 question on a 7-point Likert scale. Patients will be asked whether they would recommend the approach used to others for other discussions.
Decisional conflict scale (DCS) | Baseline (immediately following appointment); 2 weeks post appointment
  The 16 items of DCS are scored on a 0-4 scale where higher scores are reflective of uncertainty about treatment choice.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Leventakos, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials